CLINICAL TRIAL: NCT04178720
Title: Clinical Evaluation of a Daily Wear Monthly Replacement Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C010
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Refractive Errors
Keywords: Contact Lens; Daily Wear; Vision Correction
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID018869 (Experimental): Lehfilcon A contact lenses worn in both eyes at least approximately 8 hours per day and approximately 5 days per week during waking hours only. The lenses will be removed nightly for cleaning and disinfection and replaced monthly over the 3-month wear period.
  Interventions: Device: Lehfilcon A contact lenses; Device: CLEAR CARE
- Biofinity (Active Comparator): Comfilcon A contact lenses worn in both eyes at least approximately 8 hours per day and approximately 5 days per week during waking hours only. The lenses will be removed nightly for cleaning and disinfection and replaced monthly over the 3-month wear period.
  Interventions: Device: Comfilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: LID018869
  Arms: LID018869
Device: Comfilcon A contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: CooperVision® BIOFINITY®; Biofinity
  Arms: Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based system for cleaning and disinfecting silicone hydrogel contact lenses
  Other Names: CLEAR CARE® Cleaning & Disinfecting Solution

SUMMARY:
The purpose of this clinical study is to evaluate the safety and effectiveness of an investigational soft contact lens compared to a commercially available soft contact lens when worn for daily wear and replaced monthly.

DETAILED DESCRIPTION:
Subjects are expected to attend 6 study visits. The expected duration of study lens exposure is approximately 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Manifest cylinder equal to or less than 0.75 diopter (D) in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Habitually wearing Biofinity contact lenses.
* Monovision contact lens wearers.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (7):
- United States (7):
  - Alcon Investigative Site, Longwood, Florida
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Medina, Minnesota
  - Alcon Investigative Site, Granville, Ohio
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 8 investigative sites located in the US.
Pre-assignment Details: Of the 119 enrolled, 1 subject was screen failed. This reporting group includes all enrolled and dispensed subjects/eyes (118/236).
Units Other Than Participants: eyes
Groups:
- Biofinity: Comfilcon A contact lenses worn in both eyes at least approximately 8 hours per day and approximately 5 days per week during waking hours only, as randomized. Lenses were removed nightly for cleaning and disinfection and replaced monthly over the 3-month wear period.
- LID018869: Lehfilcon A contact lenses worn in both eyes at least approximately 8 hours per day and approximately 5 days per week during waking hours only, as randomized. Lenses were removed nightly for cleaning and disinfection and replaced monthly over the 3-month wear period.
Period: Overall Study
Arm/Group | Biofinity | LID018869
Started | 40; 80 eyes | 78; 156 eyes
Completed | 38; 76 eyes | 77; 154 eyes
Not Completed | 2; 4 eyes | 1; 2 eyes
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Relocation | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled and dispensed subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofinity | LID018869 | Total
Number analyzed (Participants) | 40 | 78 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (7.3) | 34.4 (7.6) | 33.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 57 | 88
  Male | 9 | 21 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 38 | 74 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 12 | 14
  White | 36 | 65 | 101
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 78 | 118

OUTCOME MEASURES:

1. Primary Outcome: Distance VA (logMAR) With Study Lenses - Completed Eyes
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Dispense, Week 1 follow-up, Week 2 follow-up, Month 1 follow-up, Month 2 follow-up, Month 3 follow-up (at least 4 hours after lens insertion at each follow-up assessment visit)
Population: This analysis population includes all enrolled and dispensed subjects/eyes that completed the study with data at corresponding in-person visit.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Biofinity: Comfilcon A contact lenses worn in both eyes at least approximately 8 hours per day and approximately 5 days per week during waking hours onl, as randomized. Lenses were removed nightly for cleaning and disinfection and replaced monthly over the 3-month wear period.
Arm/Group | Biofinity | LID018869
Number analyzed (Participants) | 38 | 77
Number analyzed (eyes) | 76 | 154
logMAR
  Dispense | -0.07 (0.06) | -0.07 (0.06)
  Week 1 follow-up: number analyzed (Participants) | 37 | 77
  Week 1 follow-up: number analyzed (eyes) | 74 | 154
  Week 1 follow-up | -0.08 (0.06) | -0.07 (0.06)
  Week 2 follow-up Snellen: number analyzed (Participants) | 38 | 76
  Week 2 follow-up Snellen: number analyzed (eyes) | 75 | 152
  Week 2 follow-up Snellen | -0.07 (0.06) | -0.07 (0.06)
  Month 1 follow-up: number analyzed (Participants) | 37 | 74
  Month 1 follow-up: number analyzed (eyes) | 74 | 148
  Month 1 follow-up | -0.07 (0.06) | -0.07 (0.06)
  Month 2 follow-up: number analyzed (Participants) | 32 | 64
  Month 2 follow-up: number analyzed (eyes) | 64 | 128
  Month 2 follow-up | -0.06 (0.06) | -0.07 (0.07)
  Month 3 follow-up: number analyzed (Participants) | 37 | 77
  Month 3 follow-up: number analyzed (eyes) | 74 | 154
  Month 3 follow-up | -0.07 (0.06) | -0.06 (0.11)

2. Primary Outcome: Distance VA (logMAR) With Study Lenses - Discontinued Eyes
Description: as for outcome 1
Time Frame: Dispense, Week 1 follow-up, Week 2 follow-up, Month 1 follow-up
Population: This analysis population includes all enrolled and dispensed subjects/eyes that discontinued the study early with data at corresponding in-person visit.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID018869
Number analyzed (Participants) | 2 | 1
Number analyzed (eyes) | 4 | 2
logMAR
  Dispense | -0.06 (0.07) | 0.00 (0.00)
  Week 1 follow-up: number analyzed (Participants) | 1 | 1
  Week 1 follow-up: number analyzed (eyes) | 2 | 2
  Week 1 follow-up | -0.12 (0.00) | -0.12 (0.00)
  Week 2 follow-up: number analyzed (Participants) | 1 | 1
  Week 2 follow-up: number analyzed (eyes) | 2 | 2
  Week 2 follow-up | 0.00 (0.00) | -0.12 (0.00)
  Month 1 follow-up: number analyzed (Participants) | 0 | 1
  Month 1 follow-up: number analyzed (eyes) | 0 | 2
  Month 1 follow-up |  | -0.12 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 3 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all enrolled and dispensed subjects.
Groups:
- Pre-treatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID018869 Ocular; LID018869 Nonocular/Systemic: Events reported in this group occurred while exposed to lehfilcon A contact lenses
- Biofinity Ocular; Biofinity Nonocular/Systemic: Events reported in this group occurred while exposed to comfilcon A contact lenses
Arm/Group | Pre-treatment | LID018869 Ocular | LID018869 Nonocular/Systemic | Biofinity Ocular | Biofinity Nonocular/Systemic
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/156 | 0/78 | 0/80 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/156 | 0/78 | 0/80 | 0/40
Other Adverse Events (participants affected / at risk) | 0/118 | 0/156 | 0/78 | 0/80 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04178720/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04178720/SAP_001.pdf